CLINICAL TRIAL: NCT06588361
Title: Examination of the Effect of Training Based on Kolcoba Comfort Theory on Dyspnea, Functional Status and Comfort Status in COPD Patients
Brief Title: Impact of Kolcaba Comfort Theory Training on Dyspnea, Function, and Comfort in COPD Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Collaborators: Scientific Research Projects Coordination Unit (Ambiguous)
Responsible Party: Principal Investigator, Şeyda Karasu, research assistant, Ataturk University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: seydakarasu
Record Dates: First submitted 2024-08-26; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Main Heading (Descriptor) Terms
Keywords: COPD; Dyspnea; Functional Status; Comfort States; Kolcaba's Comfort Theory; Education
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPD patients (Experimental): Experimental group will receive training based on Kolcaba's Comfort Theory once a week for 5 weeks.No interventions will be provided to the control group.
  Interventions: Other: Training Based on Kolcoba Comfort Theory

INTERVENTIONS:
Other: Training Based on Kolcoba Comfort Theory — Training Based on Kolcoba Comfort Theory

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is the third most fatal chronic disease worldwide, following cardiovascular diseases and cancer. COPD is characterized by chronic respiratory symptoms due to abnormalities in the airways (bronchitis/bronchiolitis) or alveoli (emphysema), leading to persistent and often progressive airway obstruction. Patients frequently experience a range of physical and psychosocial symptoms, including dyspnea, cough, sputum production, fatigue, anxiety, and depression. Dyspnea, in particular, can significantly reduce quality of life, impair daily activities, and affect patient comfort.

Functional status is a crucial metric for assessing disease progression and symptom severity in COPD and is directly related to the intensity of symptoms such as dyspnea. Effective management of symptoms and enhancement of comfort levels are critical in COPD treatment. Kolcaba's Comfort Theory provides a comprehensive approach to nursing care by addressing physical, psychospiritual, social, and environmental dimensions of patient needs. This theory can be an effective guide for improving comfort in COPD patients.

The objective of this study is to evaluate the effects of using Kolcaba's Comfort Theory as a guide in managing symptoms and enhancing the quality of care for COPD patients, focusing on dyspnea, functional status, and comfort. The research aims to provide innovative insights into the impact of Comfort Theory-based nursing care in sensitive patient populations like those with COPD and to contribute valuable information for developing effective treatment and management strategies for symptom control.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older.
* Have been diagnosed with COPD for at least 6 months.
* Be in GOLD stages 1, 2, or 3 of COPD.
* Be able to read and write in Turkish.
* Have access to a phone for communication.

Exclusion Criteria:

* Patients experiencing an acute exacerbation.
* Presence of non-COPD pulmonary problems or diagnosed cardiovascular diseases.
* Psychiatric disorders that disrupt thought processes, such as dementia or schizophrenia.
* Respiratory issues caused by diseases other than COPD.
* Problems with communication or speech.
* Use of a respiratory exercise device (PEP).
* Inability to tolerate PEP use.
* Desire to withdraw from the study at any point.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Dyspnoea-12 Scale | five monts
  It includes four Likert-type options (0=none, 1=mild, 2=moderate, 3=severe). The first seven items of the scale question the physical difficulties caused by dyspnoea in patients by evaluating whether the breath goes to all lungs, whether the patient has shortness of breath, whether there is difficulty in breathing, and whether there is effort while breathing. The remaining five items of the scale focus on the effects of breathing on emotional states such as stress, irritability, depression, distress and restlessness. The maximum score that can be obtained from the physical dimension of the scale is 21 and the maximum score that can be obtained from the emotional dimension is 15. The minimum score that can be obtained from the scale is 0 and the maximum score is 36. An increase in the score obtained from the scale indicates an increase in the severity of dyspnoea in the patient. In the original study of the scale, Cronbach's alpha value was reported as 0.90.

SECONDARY OUTCOMES:
Clinical COPD Questionnaire | five monts
  It is a questionnaire that enables the evaluation of functional status and symptoms in daily clinical practice. It consists of 10 questions questioning the last week, scored by the patient between 0-6. It consists of three areas: symptoms, mental status and functional status. The total score is calculated and divided by the number of questions, with a high score indicating a low health status (severity of COPD). The Cronbach's alpha value of the Clinical COPD Questionnaire adapted to the Turkish language was 0.90

OTHER OUTCOMES:
General Comfort Scale Short Form GCS-SF | five monts
  Its validity and reliability was performed by Sarıtaş et al. in 2018. It includes the sub-dimensions of comfort, relief (9 items), relaxation (9 items) and overcoming problems (10 items). In the evaluation of the scale consisting of positive and negative items, negative items are reverse coded and summed. The total score obtained is divided by the number of scale items and the mean value is found. The lowest possible value of 1 indicates a low comfort level and the highest value of 6 indicates a high comfort level. Reverse expressions: 2,3,7,8,8,9,10,11,12,13,14,15,16,18,20,21,23,24,25,27. The lowest possible value of 1 indicates low comfort and the highest value of 6 indicates high comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)